CLINICAL TRIAL: NCT03846284
Title: Caudal Versus Intravenous Magnesium Sulfate In The Prevention OF Emergence Agitation After Sevoflurane Anesthesia For Lower Abdominal Surgeries In Children.
Brief Title: Caudal Versus Intravenous Magnesium Sulfate on Emergence Agitation After Sevoflurane In Children.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Marwa Ibrahim Abdo, Lecturer of anesthesia and surgical intensive care- principal investigator, Mansoura University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS/17.05.159
Record Dates: First submitted 2019-02-10; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Emergence Agitation; Postoperative Pain
Keywords: Sevoflurane-; Emergence agitation; Magnesium sulfate; Children
MeSH Terms: conditions — Emergence Delirium; Pain, Postoperative | interventions — Bupivacaine; Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: , prospective, blind,controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The group allocation is concealed in sealed, opaque envelopes, which are not opened until participant consent has been obtained. The participants, their anesthetists, and staff providing postoperative care are blinded to group assignment. The drugs are prepared in equal aliquots with code numbers. Closed envelop will be used
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bupivacaine (B group) (Placebo Comparator): caudal block with bupivacaine 0.25% 1mg/kg diluted in 10 cm saline.
  + I.V injection of 10 cm saline over 10 mins then, I.V infusion 50 cm saline with rate 10-20 ml/h according to child weight.
  Interventions: Drug: Bupivacaine
- Magnesium sulfate caudal (MC group) (Experimental): caudal block with bupivacaine 0.25% 1mg/kg + Magnesium sulfate 50 mg diluted in 10 cm saline.
  + I.V injection of 10 cm saline over 10 mins then, I.V infusion of 50 cm saline with rate 10-20 ml/h according to child weight.
  Interventions: Drug: Bupivacaine; Drug: Magnesium sulfate 50mg
- Magnesium sulfate I.V (M V group) (Experimental): caudal block with bupivacaine 0.25% 1mg/kg diluted in 10 cm saline.
  + I.V injection of Magnesium sulfate 30mg/kg diluted in 10 cm saline over 10 mins then, I.V infusion one ampule of Magnesium sulfate 500mg diluted in 50 cm saline with rate 10 mg/kg/h.
  Interventions: Drug: Bupivacaine; Drug: Magnesium sulfate 30 mg

INTERVENTIONS:
Drug: Bupivacaine — caudal block with bupivacaine 0.25% 1mg/kg diluted in 10 cm saline.
  Other Names: local anesthetic drug
Drug: Magnesium sulfate 50mg — caudal block with bupivacaine 0.25% 1mg/kg plus Magnesium sulfate 50 mg diluted in 10 cm saline.
  Other Names: non anesthetic N-methyl-D-aspartate receptor antagonist
  Arms: Magnesium sulfate caudal (MC group)
Drug: Magnesium sulfate 30 mg — caudal block with bupivacaine 0.25% 1mg/kg diluted in 10 cm saline.
  + I.V injection of Magnesium sulfate 30mg/kg diluted in 10 cm saline over 10 mins then, fol I.V infusion one ampule of Magnesium sulfate 500mg diluted in 50 cm saline with rate 10 mg/kg/h.
  Other Names: non anesthetic N-methyl-D-aspartate receptor antagonist
  Arms: Magnesium sulfate I.V (M V group)

SUMMARY:
Sevoflurane is the agent of choice for induction and maintenance of day care anesthesia in children and has a wide acceptance among pediatric anesthesiologists.

Emergence agitation (EA) is a frequent postoperative complication in pediatric patients receiving inhalational anesthetics with a rapid recovery, e.g. sevoflurane Magnesium sulfate is a non anesthetic N-methyl-D-aspartate receptor antagonist, Regional anesthetic techniques have major two benefits which are lowering anesthetic requirements intraoperatively and providing adequate postoperative pain relief.

Magnesium sulfate is an adjuvant that alters the perception and duration of pain by serving as an antagonist of N-methyl-D-aspartate glutamate receptors. Caudal injection of bupivacaine with magnesium sulfate in pediatric patients after inguinoscrotal operations provided adequate postoperative analgesia without producing many side effects. Caudal block with local anesthetic with or without adjuvants may prevent emergence agitation with effective postoperative pain management.

* So the aim of this study is to compare the efficacy of caudal versus intravenous magnesium sulfate infusions in controlling emergence agitations after inhalational sevoflurane anesthesia in children who will undergo lower abdominal surgeries.

Participants and methods

All participants will receive caudal block with bupivacaine 0.25% 1mg/kg dialed in 10 cm saline.

The participants will be divided to 3 groups

1. Bupivacaine group (B group) (group 1) N = 31 :-
2. Magnesium sulfate caudal group (MC group) (group 2) N = 31 :-
3. Magnesium sulfate I.V group (MV group) (group 3) N = 31 :-

Postoperative assessment in the ( PACU):-

* The oxygen saturation (SO2), heart rate (HR), and mean arterial pressure (MAP) are monitored by the observer blinded to group allocation on admission and 10 mins till discharge (0, 10, 20, 30, 40, 50, 60mints, time of discharge) from the PACU.
* Emergence agitations (Pediatric anesthesia emergency delirium scale (PAED) The presence of Emergence agitation and its severity will be measured using (PAED).

The presence of Pain and its severity will be measured using FLACC scale.

* Time of first postoperative administration of fentanyl in mints
* Modified Aldrete score :- The discharge from the PACU will be measured using Modified Aldrete score.

DETAILED DESCRIPTION:
Participants and methods All participants will receive caudal block with bupivacaine 0.25% 1mg/kg diluted in 10 cm saline.

The participants will be divided to 3 groups

1. Bupivacaine group (B group) (group 1) N = 31 :- The participants will receive caudal block with bupivacaine 0.25% 1mg/kg diluted in 10 cm saline.

   + I.V injection of 10 cm saline over 10 mins then, followed by I.V infusion 50 cm saline with rate 10-20 ml/h according to child weight.
2. Magnesium sulfate caudal group (MC group) (group 2) N = 31 :- The participants will receive caudal block with bupivacaine 0.25% 1mg/kg plus Magnesium sulfate 50 mg diluted in 10 cm saline.

   * I.V injection of 10 cm saline over 10 mins then, followed by I.V infusion of 50 cm saline with rate 10-20 ml/h according to child weight.
3. Magnesium sulfate I.V group (MV group) (group 3) N = 31 :- The participants will receive caudal block with bupivacaine 0.25% 1mg/kg diluted in 10 cm saline.

   + I.V injection of Magnesium sulfate 30mg/kg diluted in 10 cm saline over 10 mins then, followed by I.V infusion one ampule of Magnesium sulfate 500mg diluted in 50 cm saline with rate 10 mg/kg/h.

   Standard monitoring is used during anesthesia and surgery include :- electrocardiography, non-invasive arterial pressure, arterial oxygen saturation using pulse oximeter and end-tidal concentrations are measured using capnography.

   An intravenous line is secured before induction of anesthesia, all participants will receive a standardized rapid sequence induction of anesthesia and oxygen administration for 3 minutes. Anesthesia is induced with Inhalation of 8% sevoflurane without use of muscle relaxant, cricoid pressure is applied and the trachea intubated with a suitable-size endotracheal tube. Maintained end-tidal sevoflurane concentration will be between 2.5-3.5 and will be titrated. The participants will breath spontaneously during surgery and tidal volume will be adjusted to maintain normocarbia. I.V injection of 0.2 mg/kg dexamethasone after induction as a prophylaxis of post-operative nausea and vomiting of Mg sulfate. Caudal block will be performed to participants before surgical incision with 1 of 2 investigators using the following technique :- The Participants are placed in left lateral position after induction of general anesthesia. The back of the participant including the sacral hiatus are carefully sterilized with an antiseptic solution and sterile drapes will be placed around the injection site. The technique will be done by introducing a 23-gauge hypodermic needle perpendicular to the sacrococcygeal membrane with the bevel in the direction of the long fibers of the membrane. The needle will be inserted until there is release of impedance as it pierced the sacrococcygeal membrane. Then, it is directed upwards so that it make an angle of 20-30° with the skin about 2 mm so that the whole bevel will be inside the sacral canal. The injection will be made over a period of about 60 s and then a small elastoplast dressing is placed over the injection site and the participant will be placed supine. Intraoperative analgesic supplement will not be given.

   Caudal block will be failed if HR &/or MAP increased 10 more than the previous basal value of beginning of surgery.participants will be fasting 4-6 hours for solid foods and 2 hours for clear fluids. Balanced fluid therapy containing Na Cl, glucose, K and Ca will be infused according to body weight as follows :1st 10 kg 4 ml/kg/hour, 2nd 10 kg 2 ml/kg/hour and 1 ml//hour for every 1 kg.

   Then, anesthetic gas discontinued and replaced O2 100%. At the end of the operation the trachea is extubated, The participants will be transferred to the postanesthesia care unit (PACU).

   Intraoperative assessment:-

   • Heart rate (HR) and mean arterial blood pressure (MAP), oxygen saturation (SO2) are recorded basal before operation and every 10 mins. until the end of surgery.

   • minimal alveolar concentration (MAC) of sevoflurane is recorded every 10 mins.

   • The occurrence of intraoperative hypotension (defined as systolic arterial pressure 70 plus twice the age in years and associated with altered peripheral perfusion), requiring a fluid bolus.
   * The occurrence of intraoperative bradycardia (defined as heart rate below 60 beats min for ages above 1 years), requiring atropine.
   * Duration of anesthesia: it is the time from start of inhalation induction by sevoflurane till tracheal extubation in mins.
   * Extubation time: it is the time from termination of sevoflurane to tracheal extubation in mins.
   * Emergence time: it is the time from the end of surgery till the opening of patient's eyes in mins.
   * Interaction time: it is interval between stopping sevoflurane and verbal or physical response in mins. All are noted.

   Postoperative assessment in the ( PACU):-
   * The oxygen saturation (SO2), heart rate (HR), and mean arterial pressure (MAP) are monitored by the observer blinded to group allocation on admission and 10 mins till discharge (0, 10, 20, 30, 40, 50, 60mints, time of discharge) from the PACU.
   * Emergence agitations (Pediatric anesthesia emergency delirium scale (PAED):- The presence of Emergence agitation and its severity will be measured using (PAED).

   Item 1. The participant makes eye contact with care giver 2. The child's actions are purposeful 3. The child is aware of his/her surroundings 4. The child is restless 5. The child is inconsolable - Items 1, 2 and 3 are scored: 4 = not at all, 3 = just a little, 2 quite a bit, 1 = very much, 0 = extremely.

   - Items 4 and 5 are scored: 0 = not at all, 1 = just a little, 2 = quite a bit, 3 = very much, 4 = extremely.

   It will be monitored on admission and every 10 mins till discharge from the PACU (0, 10, 20, 30, 40, 50, 60 mins, time of discharge).

   PAED score ≥ 10 will be managed by intravenous doses of fentanyl 1micg/kg, repeated after 10 min if the child is still agitated, with a maximum total dose of 2 micg/kg. (PAED) score ≥ 10 will be considered to be a diagnostic endpoint for the development of agitation.

   • Pain score (FLACC scale) :-

   The presence of Pain and its severity will be measured using FLACC scale.

   CATEGORIES SCORING

0 1 2 Face

No particular expression or smile Occasional grimace or frown, withdrawn, disinterested. Frequent to constant quivering chin, clenched jaw. Legs

Normal position or relaxed. Uneasy, restless, tense. Kicking, or legs drawn up.

ACTIVITY

Lying quietly, normal position moves easily Squirming, shifting back and forth, tense. Arched, rigid or jerking. Cry

No cry, (awake or asleep) Moans or whimpers;occasional complaint crying steadily, screams or sobs, CONSOLABILITY

Content, relaxed. Reassured by occasional touching hugging or being talked to, distractable. Difficulty to console or comfort

It will be monitored on admission and every 10 mins till discharge from the PACU (0, 10, 20, 30, 40, 50, 60 mins, time of discharge). If the FLACC pain scale score is noted at any time to be 4 or more, the patient will be given1micg/kg fentanyl I.V and repeated after 10 mins, if the participant is still in pain with a maximum total dose 2 mg/kg

* Time of first postoperative administration of fentanyl :- in mints
* Modified Aldrete score :- The discharge from the PACU will be measured using Modified Aldrete score. Items are :-

Activity:

2. able to move 4 extremities voluntarily or on command

1. able to move 2 extremities voluntarily or on command 0. unable to move extremities voluntarily or on command

Respiration:

2. able to breath deeply and cough freely

1. dyspnea or limited breathing 0. apneic

Circulation:

2. BP +/- 20% of pre-anesthetic level

1. BP +/- 20% to 49% of pre-anesthetic level 0. BP +/- 50% of pre-anesthetic level

Consciousness:

2. fully awake

1. arousable on calling 0. not responding

O2 saturation :

2. able to maintain O2 saturation <92% on room air

1. needs O2 inhalation to maintain O2 saturation <90% 0. O2 saturation >90% even with O2 supplement. It will be monitored on admission and every 10 mins till discharge from the PACU (0, 10, 20, 30, 40, 50, 60 mins, time of discharge). Participants will be discharged from the PACU after adequate control of agitation and pain, and when they has achieved Modified Aldrete score characteristics of ≥ 9,

Postoperative complications :- All post operative complications are also recorded by the observer blinded to group allocation which include :-

* The occurrence of Postoperative nausea and vomiting (PONV) :-
* (PONV) is treated as needed with i.v.ondansetron 0.06 mg/kg every 4 h.
* The occurrence of postoperative respiratory depression (defined as oxygen saturation below than 95%) and respiratory rate below than 10 breaths/min.
* The occurrence of Postoperative Laryngospasm or Bronchospasm.
* The occurrence of postoperative Hypotension definition and treatment as mentioned before.
* The occurrence of postoperative Bradycardia definition and treatment as mentioned before.

Statistical analysis

Statistical analysis will be done by using statistical package for social scientists (SPSS) program version 16. Data will be proved parametric by using kolmogorov -Smi mov test. The quantitative data will be presented in the form of mean and standard Deviation. One-way ANOVA test will be used to compare between quantitative data of the three groups. Paired t-test will be used to study between two values in the same group. Pain score, sedation score will be represented by median and range and will be analyzed by Kruskal-Wallis test to compare between the three groups. Mann-Whitney test will be used for comparison between 2 groups separately. Significance will be considered when P-value is less than 0.05

Sample size The primary outcomes was the incidence of emergence agitation. A previous study on the effect of magnesium sulfate infusion on the incidence and severity of emergence agitation in children under going adenotonsillectomy under sevoflurane anesthesia reported a 72% incidence of emergence agitation. (14). We presumed that a clinically significant difference would be 50% between the incidence of agitation in the intervention and control groups. With a power of 85% (a = 0.05, two-tailed), the sample size was calculated to be 93 patients (31 in each group). The sample size was calculated using Power Analysis and Sample Size 12 software (NCSS, Kay seville, ut USA).

ELIGIBILITY:
Inclusion Criteria:

-All participants undergoing lower abdominal surgeries

Exclusion Criteria:

All participants with:-

* history of developmental delay,
* mental retardation,
* psychological disorders or
* Epilepsy which can make observational pain intensity assessment difficult,
* a known or suspect coagulopathy,
* a known allergy to any of the study drugs and
* any signs of infection at the site of the proposed caudal block.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2017-10-08 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With sevoflurane-agitation are Assessed by Pediatric anesthesia emergency delirium scale (PAED) in 3 groups caudal versus intravenous magnesium sulfate infusions or caudal block alone | up to 96 weeks
  (PAED).
  1. The child makes eye contact with care giver
  2. The child's actions are purposeful
  3. The child is aware of his/her surroundings
  4. The child is restless
  5. The child is inconsolable
     * Items 1, 2 and 3 are scored: 4 = not at all, 3 = just a little, 2 quite a bit, 1 = very much, 0 = extremely.
     * Items 4 and 5 are scored: 0 = not at all, 1 = just a little, 2 = quite a bit, 3 = very much, 4 = extremely.
     * minimal score 0 maximal score 20
     * It will be monitored on admission and every 10 mins till discharge from the PACU (0, 10, 20, 30, 40, 50, 60 mins, time of discharge).
  PAED score ≥ 10 fentanyl 1micg/kg I V will be given, repeated after 10 min if still agitated, with a maximum total dose of 2 micg/kg. (PAED) score ≥ 10 will be considered to be a diagnostic endpoint for agitation.

SECONDARY OUTCOMES:
Number of Participants With Pain and its severity will be measured using FLACC in 3 groups caudal versus intravenous magnesium sulfate infusions or caudal block alone after inhalational sevoflurane anesthesia in children | up to 96 weeks
  FLACC scale
  0 1 2 Face No expression Occasional grimace , . Frequent quivering chin, clenched jaw.
  Legs Normal position . Uneasy,. legs drawn up. Activity Lying quietly. shifting back . Arched, rigid . Cry No cry whimpers; Crying steadily, screams, Consolability Content, . Reassured by being talked to, . Difficulty to console
  * It will be monitored on admission and every 10 mins till discharge from the (0, 10post anesthetic care unit, 20, 30, 40, 50, 60 mins, time of discharge).
  * minimal score is 0.maximal score is 12
  * If the FLACC pain scale score is noted at any time to be 4 or more, 1micg/kg fentanyl I.V and repeated after 10 mins, will be given
  -Time of first postoperative administration of fentanyl in mints -
The discharge from the post anesthetic care unit will be measured using Modified Aldrete score after inhalational sevoflurane anesthesia in children in 3 groups | up to 96 weeks
  Modified Aldrete score
  Activity:
  2. able to move 4 extremities
  1. able to move 2 extremities 0. unable to move extremities
  Respiration:
  2. able to breath deeply
  1. dyspnea 0. apneic
  Circulation:
  2. BP +/- 20% of pre-anesthetic level
  1. BP +/- 49% 0. BP +/- 50%
  Consciousness:
  2. fully awake
  1. arousable on calling 0. not responding
  O2 saturation :
  2. O2 saturation <92% on room air
  1. needs O2 O2 saturation <90% 0. O2 saturation >90%
  * It will be monitored on admission and every 10 mins till discharge from the PACU (0, 10, 20, 30, 40, 50, 60 mins, time of discharge).
  * minimal score is 0 maximal score is 10
  * Patients will be discharged from post anesthetic care unit after adequate control of agitation and pain, and when they has achieved Modified Aldrete score characteristics of ≥ 9,

CONTACTS AND LOCATIONS:
Overall Officials: Gehan Ad Tarabeah, MD, Study Chair — Profosser of anesthesia and surgical intensive care; Hesham Ah Abdel Mohaiemn, MD, Study Director — Assisstant professor of anesthesia and surgical intensive care; Marwa Ib Abdo, MD, Study Director — Lecturer of anesthesia and surgical intensive care; Mahmoud Mo Abdel latef, Ph.D, Principal Investigator — Resident of anesthesia and surgical intensive care
Locations (1):
- Marwa ibrahim mohamed abdo, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tomal CR, Silva AG, Yamashita AM, Andrade PV, Hirano MT, Tardelli MA, Silva HC. Assessment of induction, recovery, agitation upon awakening, and consumption with the use of two brands of sevoflurane for ambulatory anesthesia. Rev Bras Anestesiol. 2012 Mar-Apr;62(2):154-72. doi: 10.1016/S0034-7094(12)70115-0. PMID 22440372
- [Background] Dahmani S, Stany I, Brasher C, Lejeune C, Bruneau B, Wood C, Nivoche Y, Constant I, Murat I. Pharmacological prevention of sevoflurane- and desflurane-related emergence agitation in children: a meta-analysis of published studies. Br J Anaesth. 2010 Feb;104(2):216-23. doi: 10.1093/bja/aep376. Epub 2010 Jan 3. PMID 20047899
- [Background] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210
- [Background] Ahuja S, Aggarwal M, Joshi N, Chaudhry S, Madhu SV. Efficacy of Caudal Clonidine and Fentanyl on Analgesia, Neuroendocrine Stress Response and Emergence Agitation in Children Undergoing Lower Abdominal Surgeries Under General Anaesthesia with Sevoflurane. J Clin Diagn Res. 2015 Sep;9(9):UC01-5. doi: 10.7860/JCDR/2015/12993.6423. Epub 2015 Sep 1. PMID 26500980
- [Background] Patel A, Davidson M, Tran MC, Quraishi H, Schoenberg C, Sant M, Lin A, Sun X. Dexmedetomidine infusion for analgesia and prevention of emergence agitation in children with obstructive sleep apnea syndrome undergoing tonsillectomy and adenoidectomy. Anesth Analg. 2010 Oct;111(4):1004-10. doi: 10.1213/ANE.0b013e3181ee82fa. Epub 2010 Aug 12. PMID 20705788
- [Background] Silva LM, Braz LG, Modolo NS. Emergence agitation in pediatric anesthesia: current features. J Pediatr (Rio J). 2008 Mar-Apr;84(2):107-13. doi: 10.2223/JPED.1763. PMID 18372935
- [Background] Kim MS, Moon BE, Kim H, Lee JR. Comparison of propofol and fentanyl administered at the end of anaesthesia for prevention of emergence agitation after sevoflurane anaesthesia in children. Br J Anaesth. 2013 Feb;110(2):274-80. doi: 10.1093/bja/aes382. Epub 2012 Oct 26. PMID 23103775
- [Background] Albrecht E, Kirkham KR, Liu SS, Brull R. Peri-operative intravenous administration of magnesium sulphate and postoperative pain: a meta-analysis. Anaesthesia. 2013 Jan;68(1):79-90. doi: 10.1111/j.1365-2044.2012.07335.x. Epub 2012 Nov 1. PMID 23121612
- [Background] Abdulatif M, Ahmed A, Mukhtar A, Badawy S. The effect of magnesium sulphate infusion on the incidence and severity of emergence agitation in children undergoing adenotonsillectomy using sevoflurane anaesthesia. Anaesthesia. 2013 Oct;68(10):1045-52. doi: 10.1111/anae.12380. Epub 2013 Aug 3. PMID 23909742
- [Background] Stewart DW, Ragg PG, Sheppard S, Chalkiadis GA. The severity and duration of postoperative pain and analgesia requirements in children after tonsillectomy, orchidopexy, or inguinal hernia repair. Paediatr Anaesth. 2012 Feb;22(2):136-43. doi: 10.1111/j.1460-9592.2011.03713.x. Epub 2011 Oct 25. PMID 22023485
- [Background] Farrag WS, Ibrahim AS, Mostafa MG, Kurkar A, Elderwy AA. Ketamine versus magnesium sulfate with caudal bupivacaine block in pediatric inguinoscrotal surgery: A prospective randomized observer-blinded study. Urol Ann. 2015 Jul-Sep;7(3):325-9. doi: 10.4103/0974-7796.152039. PMID 26229319
- [Background] Benzon HA, Shah RD, Hansen J, Hajduk J, Billings KR, De Oliveira GS Jr, Suresh S. The Effect of Systemic Magnesium on Postsurgical Pain in Children Undergoing Tonsillectomies: A Double-Blinded, Randomized, Placebo-Controlled Trial. Anesth Analg. 2015 Dec;121(6):1627-31. doi: 10.1213/ANE.0000000000001028. PMID 26501831
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Aldrete JA. The post-anesthesia recovery score revisited. J Clin Anesth. 1995 Feb;7(1):89-91. doi: 10.1016/0952-8180(94)00001-k. No abstract available. PMID 7772368